CLINICAL TRIAL: NCT04749719
Title: At Home Brain Stimulation Studies of Memory and Memory Awareness
Acronym: remTDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooklyn College of the City University of New York (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Chua, Associate Professor, Brooklyn College of the City University of New York
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 42037; SC3GM121192 (NIH)
Record Dates: First submitted 2021-02-01; First posted 2021-02-11 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation; memory; metacognition; brain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DLPFC stimulation (Experimental): F3-SO montage or OLE optimized with 2 mA stimulation for up to 30 min during memory and metamemory task.
  Interventions: Device: remotely supervised transcranial direct current stimulation
- Sham tDCS (Sham Comparator): F3-SO montage or OLE optimized with sham stimulation for up to 30 min during memory and metamemory task.
  Interventions: Device: remotely supervised transcranial direct current stimulation

INTERVENTIONS:
Device: remotely supervised transcranial direct current stimulation — Low levels of electrical current are applied across the scalp to induce small changes in brain activity. This is done using remote supervision.

SUMMARY:
The main goal of this research is to determine the role of several brain regions in memory processes and cognitive functions. Participants will be remotely supervised via video chat while self-administering tDCS, a form of non-invasive brain stimulation. Before participating in the experiment, participants will be properly trained on use of the remote tDCS device and screened for eligibility. While using the tDCS device, participants will be engaging in tasks that assess different aspects of memory and executive functioning. By using remotely supervised tDCS while participants are completing these cognitive tasks, we will be able to make causal claims about the role of the targeted brain regions in different cognitive processes.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-35
* normal or corrected to normal vision
* fluent in English and speaking English since age 5
* right handed

Exclusion Criteria:

* chronic skin disease or medical skin condition
* unhealed wound or open skin on the scalp, face, neck, or forehead
* metal or electrode implants (e.g., cochlear implants, pacemakers, metal plates, rods, or screws in their head; for complete detail, see the screening form)
* seizures or a family history of seizures, or are taking medications with a lowered seizure threshold
* pregnant or lactating
* any neurologic or psychiatric diseases
* certain hair styles (dreadlocks, cornrows, etc) or hair coverings (e.g., wigs, hajibs, etc that will not be removed; note that a request can be made for an experimenter of a specific gender)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-21 (Estimated)

PRIMARY OUTCOMES:
Memory performance | through study completion, an average of 4 weeks
  % Correct on the Memory Task

SECONDARY OUTCOMES:
Memory Confidence | through study completion, an average of 4 weeks
  Average % Confidence on the Memory Task

OTHER OUTCOMES:
Metamemory Accuracy | through study completion, an average of 4 weeks
  Calibration and resolution of confidence and accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooklyn College, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No